CLINICAL TRIAL: NCT03360396
Title: A Randomized Controlled Study of PneumRx Endobronchial Coil System Versus Standard-of-Care Medical Management in the Treatment of Subjects With Severe Emphysema
Brief Title: Study of PneumRx Endobronchial Coil System in Treatment of Subjects With Severe Emphysema
Acronym: ELEVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTG-004517-01
Record Dates: First submitted 2017-11-22; First posted 2017-12-04 (Actual); Results first posted 2021-11-03 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Emphysema
Keywords: severe heterogeneous emphysema; severe homogeneous emphysema
MeSH Terms: conditions — Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Endobronchial Coils (Experimental): Treatment with PneumRx Endobronchial Coil System
  Interventions: Device: Endobronchial Coils
- Control (No Intervention): Medically-managed control group

INTERVENTIONS:
Device: Endobronchial Coils — Endobronchial Coil implants
  Arms: Endobronchial Coils

SUMMARY:
This study will look at outcomes between Endobronchial Coil Treatment and Control groups in patients with severe heterogeneous and or homogeneous emphysema.

DETAILED DESCRIPTION:
This will be a prospective, multicenter, randomized, controlled study comparing outcomes between the Endobronchial Coil and Control Groups. Subjects will be block randomized in a Treatment to Control ratio of 2:1. The randomization will be stratified by site and homogeneous versus heterogeneous emphysema, to support a balance of patients with differing heterogeneity in both the Treatment and Control Groups

ELIGIBILITY:
Inclusion Criteria:

* Read, understood and signed the Informed Consent form
* Meets indications for use per the IFU
* Bilateral heterogeneous and/or homogeneous emphysema
* Post bronchodilator 15% predicted ≤ Forced Expiratory Volume in 1 second (FEV1) ≤ 45% predicted
* Post bronchodilator Residual Volume (RV) ≥ 200% predicted
* Post bronchodilator Total Lung Capacity (TLC) >100% pred.
* Post bronchodilator RV/TLC > 55%
* Dyspnea related to hyperinflation scored ≥ 2 on modified Medical Research Council (mMRC) dyspnea scale despite optimal medical management
* Receiving optimal drug therapy and medical management according to clinical practice.
* Performing regular physical activity, at least 2 times per week
* Stopped smoking as confirmed by carboxyhemoglobin (CoHB)
* 100m ≤ 6 minute walk distance (6MWD) ≤ 450m
* Deemed eligible per Eligibility Review Committee (ERC)
* if treated in France, subject must be entitled to French social security.

Exclusion Criteria:

* Known sensitivity to drugs required for performing bronchoscopy or in whom bronchoscopic procedures are contraindicated
* Evidence of active infection in the lungs
* Hypersensitivity or allergy to nitinol (nickel-titanium) or its constituent metals
* Clinical significant pulmonary fibrosis
* Clinically significant, generalized bronchiectasis
* Clinically significant bleeding disorders
* Patient taking immunosuppressive drugs other than steroids (e.g., for the treatment of cancer, rheumatoid arthritis, autoimmune disease, or prevention of tissue or organ rejection).
* Primary diagnosis of asthma
* Two (2) or more COPD exacerbations in the prior year, or 1 or more COPD exacerbations in the prior 3 months with indication for hospitalization assessment, according to GOLD 2017 recommendations .
* Predominant small airways disease defined as significant bronchiectasis with sputum production (> 2 tablespoons daily) or significant bronchial wall thickening per High Resolution Computed Tomography (HRCT)
* Percent Low Attenuation Area (%LAA) < 20% in the most damaged lobe of either lung.
* Computed Tomography (CT) Imaging consistent with active pulmonary infection, significant interstitial disease or pleural disease
* Severe bullous disease (defined by bulla > 8cm or 1/3 of lung volume, or single bullous defect >8 cm) or predominant paraseptal emphysema [defined by numerous large (>1cm) paraseptal defects in the target lobe comprising of >5% of total lung volume].
* Lung pathology of nodule not proven stable or benign
* Radiographic confirmation of atelectasis or other scarring/fibrosis in areas of intended Coil implant
* Use of more than 20 mg/day prednisolone or equivalent dosage of a different corticosteroid
* Severe pulmonary hypertension (Right Ventricular Systolic Pressure (RVSP) > 50 mm Hg or other signs of Pulmonary Hypertension (PHT) with right ventricular dysfunction)
* Severe hypercapnia (PaCO2 > 55 mmHg on room air) and/or severe hypoxemia (PaO2 < 45mm Hg on room air, High altitude criterion: PaO2 < 30 mm Hg)
* Previous Lung Volume Reduction (LVR) surgery, lung transplantation, lobectomy, LVR devices or other device to treat COPD in either lung.
* Diagnosed with alpha-1 antitrypsin deficiency
* Diffusion Capacity of the lungs for Carbon Monoxide (DLCO) < 20 %
* Significant, recent or unstable cardiac disease defined as severe heart failure (Left Ventricular Ejection Fraction (LVEF) < 45% despite optimal medical management), unstable cardiac arrhythmia or coronary artery disease (angina on activity), or ischemic event in the past 6 months.
* Body Mass Index (BMI) > 30
* Participation in any other clinical Study.
* Subject is pregnant or lactating, or plan to become pregnant within the study timeframe.
* If treated in France, Subject is a "personnel vulnerable" as defined by French Regulation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix Herth, MD,, Principal Investigator — University Hospital Heidelberg; Arschang Valipour, MD,FCCP,PhD, Principal Investigator — Nord-Klinik Floridsdorf
Locations (19):
- Ludwig Boltzmann Institut Fur COPD und pneumologische Epidemologie, Vienna, Austria
- France (6):
  - CHU Grenoble, Grenoble
  - CHU Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nice, Nice
  - Hôpital Bichat, Paris
  - CHU de Reims - Hopital Maison Blanche, Reims
  - Nouvel Hôpital Civil, Strasbourg
- Germany (9):
  - Charite Berlin - Medizinische Klinik mit Schwerpunkt Infektiologie und Pneumologie, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe GmbH, Berlin
  - Universitätsklinkum Bonn, Bonn
  - Ruhrlandklinik Essen, Essen
  - Thoraxklinik, Heidelberg
  - Lungenklinik, Hemer
  - Lungenfachklinik Immenhausen, Immenhausen
  - Klinikverbund Kempten-Oberallgäu, Immenstädt
  - Krankenhaus vom Roten Kreuz Bad Cannstatt GmbH, Stuttgart
- Ospedale Careggi, Florence, Italy
- University Medical Center Groningen, Groningen, Netherlands
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agrawal A. Interventional Pulmonology: Diagnostic and Therapeutic Advances in Bronchoscopy. Am J Ther. 2021 Feb 9;28(2):e204-e216. doi: 10.1097/MJT.0000000000001344. PMID 33590989

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endobronchial Coils | Control
Started | 80 | 40
Completed | 0 | 0
Not Completed | 80 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endobronchial Coils | Control | Total
Number analyzed (Participants) | 80 | 40 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (7.51) | 62.8 (7.06) | 63.2 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 21 | 62
  Male | 39 | 19 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 78 | 40 | 118
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: Litres] | 0.8 (0.2026) | 0.8 (0.2220) | 0.8 (0.21)
St. George Respiratory Questionnaire Score (SGRQ) [Mean (Standard Deviation); unit: units on a scale] | 59.327 (11.4232) | 54.666 (14.5222) | 57.8 (12.67)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in FEV1 at 6 Months
Description: Percent change in FEV1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Endobronchial Coils | Control
Number analyzed (Participants) | 57 | 34
percent change from baseline | 12.745 (33.1782) | -2.604 (10.1628)
Statistical Analysis 1: Comparison: Endobronchial Coils vs Control; Study was closed early in all regions except for France. Statistical Analysis plan was updated to include descriptive statistics only. Sites in France remain open and all subjects in France will be followed through 36 months; Test type: Other — Study was closed early in all regions except for France. Statistical Analysis plan was updated to include descriptive statistics only. Sites in France remain open and all subjects in France will be followed through 36 months; Study was closed early in all regions except for France. Statistical Analysis plan was updated to include descriptive statistics only. Sites in France remain open and all subjects in France will be followed through 36 months; Study was closed early in all regions except for France. SAP was updated to include descriptive statistics only. French sites remain open; Study was closed early in all regions except for France. Statistical Analysis plan was updated to include descriptive statistics only. Sites in France remain open and all subjects in France will be followed through 36 months

2. Primary Outcome: Absolute Change in SGRQ Score at 6 Months
Description: Change in SGRQ score - St. George Respiratory Questionnaire from 0 to 100, higher score indicating more limitations (worse), increase in score indicating worse outcome, decrease in score indicating improvement
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Endobronchial Coils | Control
Number analyzed (Participants) | 54 | 33
score on a scale | -8.561 (14.6834) | 2.080 (9.8483)
Statistical Analysis 1: Comparison: Endobronchial Coils vs Control; Study was terminated early, and Statistical Analysis plan was updated to include descriptive statistics only; Test type: Other — Study was terminated early, and Statistical Analysis plan was updated to include descriptive statistics only; Study was terminated early, and Statistical Analysis plan was updated to include descriptive statistics only; Study was terminated early, and Statistical Analysis plan was updated to include descriptive statistics only; Study was terminated early, and Statistical Analysis plan was updated to include descriptive statistics only

3. Post Hoc Outcome: 36 Month Follow Up Visit Completion for French Participants (N=46)
Description: Number of French participants who received treatment with Endobronchial Coil System (randomized and crossover participants) that completed the 36 month follow up visit. All control participants who exited after 6 months are excluded for this outcome.
Time Frame: 36 months
Population: Global study was terminated early; however, French Authorities required French participants to be followed through 36-months for safety only. Only subjects that received treatment with Endobronchial Coil System (randomized and crossover control participants) are included in this outcome.
Measure: Number; unit: participants
Arm/Group | Endobronchial Coils | Control
Number analyzed (Participants) | 46 | 0
participants | 17 |

4. Post Hoc Outcome: Crude Mortality for French Participants (N=46)
Description: Number of deaths for French participants through 36 months. All control participants who exited after 6 months are excluded for this outcome.
Time Frame: 36 months
Population: Global study was terminated early; however, French Authorities required French participants to be followed through 36-months for safety only.
Measure: Count of Participants; unit: Participants
Arm/Group | Endobronchial Coils | Control
Number analyzed (Participants) | 46 | 0
Participants | 5 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Endobronchial Coils | Control
All-Cause Mortality (participants affected / at risk) | 5/73 | 0/40
Serious Adverse Events (participants affected / at risk) | 30/73 | 3/40
Other Adverse Events (participants affected / at risk) | 39/73 | 12/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endobronchial Coils (N=73) | Control (N=40)
Pneumonia (Infections and infestations) | 8 (8) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
urosepsis (Infections and infestations) | 1 (1) | 0 (0)
infective exacerbation of COPD (Infections and infestations) | 0 (0) | 1 (1)
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dypsnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
death (General disorders) | 1 (1) | 0 (0)
road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
device dislocation (Product Issues) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endobronchial Coils (N=73) | Control (N=40)
Ear Haemorrhage (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Gastrointestinal Tract Irritation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 10 (12) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
bronchitis (Infections and infestations) | 8 (9) | 4 (4)
Escherichia Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Infected Dermal Cyst (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (11) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT03360396/Prot_SAP_000.pdf